CLINICAL TRIAL: NCT04857255
Title: Technology-assisted Language Intervention for Children Who Are Deaf/Hard-of-hearing (TALI)
Brief Title: Technology-assisted Language Intervention (TALI)
Acronym: TALI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01DC018550 (NIH)
Record Dates: First submitted 2021-04-19; First posted 2021-04-23 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Hearing Loss, Bilateral; Language Development
Keywords: hearing loss; randomized clinical trial; intervention; language development
MeSH Terms: conditions — Hearing Loss, Bilateral; Hearing Loss | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Technology Assisted Language Intervention (TALI) (Active Comparator): Augmentative and alternative communication software incorporated into active speech-language therapy
  Interventions: Behavioral: Technology assisted language intervention
- Treatment as Usual (Active Comparator): Speech language therapy child is typically receiving (no change to current care)
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Technology assisted language intervention — speech language therapy that has integrated technology delivered through specific software on an iPad
  Arms: Technology Assisted Language Intervention (TALI)
Behavioral: Treatment as usual — No change will occur to the current ongoing speech-language therapy being delivered.
  Arms: Treatment as Usual

SUMMARY:
This study is testing the effectiveness of augmentative and alternative communication technology among deaf or hard of hearing children for improving language development. Children will be randomized to receive either the technology intervention or treatment as usual

ELIGIBILITY:
Inclusion Criteria:

* Age 3-10 years
* Documented permanent bilateral hearing loss with severity levels clinically defined moderate to profound).
* Identified with a language deficit, defined by either the ratio of language standard scores to nonverbal intelligence quotient <.85 or a differences in nonverbal IQ and language standard scores of 10 points. Language scores may either be receptive or expressive.
* Currently receiving speech-language therapy.

Exclusion Criteria:

Mild hearing loss and unilateral hearing loss

* primary language other than English
* significant motor impairments
* nonverbal IQ <80
* children with severe communication disorders (i.e. autism spectrum disorders).

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 114 (Estimated)
Dates: Start 2020-10-15 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Mean Length of Utterance in morphemes | 24 weeks
  Measurement of syntax
Mean Turn Length | 24 weeks
  Measurement of discourse
Number of different vocabulary words spoken | 24 weeks
  measure of semantics
Clinical Evaluation of Language Fundamentals-5th edition | 24 weeks
  Provides receptive and expressive standard scores on a scale with a mean of 100 +/- 15standard deviations; higher scores indicate better/higher language skills

SECONDARY OUTCOMES:
Expressive Vocabulary Test 2nd edition | 24 weeks
  Provides expressive vocabulary standard scores on a scale with a mean of 100 +/- 15standard deviations; higher scores indicate better/higher vocabulary skills
Clinical Evaluation of Language Fundamentals-5th edition-pragmatics profile | 24 weeks
  Provides pragmatic language scores as scaled scores (ranging from 1 to 15), age equivalents and percentile ranks

CONTACTS AND LOCATIONS:
Overall Officials: Jareen Meinzen-Derr, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (2):
- United States (2):
  - Children's Hospital of Colorado, Aurora, Colorado
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

DOCUMENTS (1):
  • Informed Consent Form (2021-11-06): https://cdn.clinicaltrials.gov/large-docs/55/NCT04857255/ICF_000.pdf